CLINICAL TRIAL: NCT01641393
Title: A Randomised, Double-Blind, Active-Controlled, Two-Treatment, Crossover, Multinational, Multicentre Study to Compare Two Pancreatic Enzyme Products in the Treatment of Exocrine Pancreatic Insufficiency in Subjects With Cystic Fibrosis
Brief Title: Safety and Efficacy Study of 2 Pancreatic Enzymes for Treatment of Exocrine Pancreatic Insufficiency in Cystic Fibrosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-005; 2009-012842-21 (EudraCT Number)
Record Dates: First submitted 2012-07-10; First posted 2012-07-16 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Exocrine Pancreatic Insufficiency: Cystic Fibrosis
Keywords: Exocrine Pancreatic Insufficiency; Cystic Fibrosis; Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUR-1008 then Kreon (Experimental): * EUR-1008 during Treatment Period 1 (29 days ±2 days) and
  * Kreon during Treatment Period 2 (29 days ±2 days).
  Interventions: Drug: EUR-1008 25,000 Units; Drug: Kreon 25,000 Units
- Kreon then EUR-1008 (Experimental): * Kreon during Treatment Period 1 (29 days ±2 days) and
  * EUR-1008 during Treatment Period 2 (29 days ±2 days).
  Interventions: Drug: EUR-1008 25,000 Units; Drug: Kreon 25,000 Units

INTERVENTIONS:
Drug: EUR-1008 25,000 Units — EUR-1008 25,000 Units is a PEP with pancreas powder as the active ingredient.18 Pancreas powder contains various enzymes having proteolytic, lipolytic, and amylolytic activity. Each capsule contains approximately 25,000 Ph. Eur. lipase units. EUR-1008 25,000 consists of orally administered capsules containing enteric-coated beads.
  Other Names: Zenpep
Drug: Kreon 25,000 Units — Kreon 25,000 is a PEP consisting of porcine-derived pancreatic enzymes.18 Each capsule contains approximately 25,000 Ph. Eur. lipase units. Kreon 25,000 consists of orally administered capsules containing enteric-coated spheres.
  Other Names: Kreon

SUMMARY:
The purpose of the study is to further evaluate the safety and efficacy of EUR-1008 as compared to Kreon® in the treatment of exocrine pancreatic insufficiency associated with Cystic Fibrosis in subjects 12 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

1. Definitive diagnosis of CF based on the following:

   * One clinical feature consistent with CF and
   * Either a genotype with 2 identifiable mutations known to cause CF or a sweat chloride concentration >60 mEq/L by pilocarpine iontophoresis
2. Pancreatic insufficiency documented by a monoclonal faecal elastase (FE) 100 μg/g stool at screening (test results within the previous 12 months are acceptable)
3. Currently receiving pancreatic enzyme replacement therapy
4. Adequate nutritional status based on the following: body mass index (BMI) >19 kg/m2 in adult subjects or a BMI percentile 10th percentile for age in adolescent (12 to 17 years age group) subjects
5. Are clinically stable with no evidence of concomitant illness or acute upper or lower respiratory tract infection that requires antibiotics during the 7-day interval prior to screening and preceding entry into this clinical study

Exclusion Criteria:

1. Age <12 years
2. Known contraindication, hypersensitivity, or intolerance to pork or other porcine PEPs
3. Current uncontrolled diabetes mellitus
4. History of solid organ transplantation
5. History of surgery affecting the bowel function and weight gain

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Coefficient of Fat Absorption over 72 hours (CFA-72h) | 72 hours
  During the last 72 hours of each treatment period, the CFA-72h will be calculated using fat intake data from the diet and fat excretion data from stools. Fat intake will be calculated by the dietician in collaboration with the study investigator using a validated tool.

SECONDARY OUTCOMES:
Body weight | 58 days.
  Body weight at baseline (Visit 2 [Day 0]) and at the end of each treatment period.
Coefficient of nitrogen absorption | 72 hours
  Coefficient of nitrogen absorption at the end of each treatment period as assessed by a specialised central laboratory by means of Dumas combustion method.
Control of signs and symptoms of EPI | 2- 14 day periods
  Control of signs and symptoms of EPI (as recorded in subject diaries). The following will be captured:
  * Stools frequency (number/day)
  * Stools consistency (hard, formed/normal; soft, watery, overt diarrhoea)
  * Fat or grease visible in stools (Yes/No)
  * Abdominal pain (mild, moderate, severe)
  * Bloating (mild, moderate, severe)
  * Flatulence (mild, moderate, severe)
Impact on overall health, daily life, perceived well-being, and symptoms | 58 days
  Impact on overall health, daily life, perceived well-being, and symptoms evaluated using the CFQ (administered by designated study personnel prior to randomisation and at the end of each treatment period).
Total cholesterol, calculated LDL-C, HDL-C | 58 days
  Total cholesterol, calculated LDL-C, HDL-C (sampling performed prior to randomisation and at the end of each treatment period).
Treatment Emergent Adverse Events | 78 days
  Frequency, duration, and severity of treatment-emergent adverse events (TEAEs);
Standard safety laboratory tests | 58 days
  Standard safety laboratory tests, analysed by central laboratory:
  * Haematology: red blood cell count, haemoglobin, haematocrit, total leukocytes with diff count, and platelets
  * Serum biochemistry: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total protein, albumin, total bilirubin, direct and indirect bilirubin, blood urea nitrogen, uric acid, creatinine, fasting plasma glucose, fasting cholesterol evaluations (total cholesterol, LDL-C, HDL-C, and triglycerides), fat-soluble vitamins (A, D, and E) and serum electrolytes
Vital signs | 78 days
  Vital signs including blood pressure, heart rate, respirations and body temperature.
Fat-soluble vitamins A, D, and E | 58 days
  Fat-soluble vitamins A, D, and E (sampling performed prior to randomisation and at the end of each treatment period).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Taylor, MD, PhD, Principal Investigator — Sheffield Children's Hospital, The Academic Unit of Child Health
Locations (37):
- Belgium (2):
  - University Hospital Antwerp - Universitair Ziekenhuis Antwerpen (UZA), Antwerp
  - Universitair Ziekenhuis Gent, Centrum voor Mucoviscidose, Ghent
- Bulgaria (4):
  - Clinic of Paediatric Diseases at UMHAT Dr Georgi Stranski, Pleven
  - Clinic of Genetic and Paediatric Diseases at UMHAT Sveti Georgi, Plovdiv
  - Specialized Hospital for Active Treatment of Pulmological and Phtisiatric Disease, Rousse
  - Multiprofile Clinic for Specialized Pediatric Clinic at MHAT Sveta Marina, Varna
- France (2):
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Nouvel Hôpital Civil, Strasbourg
- Germany (7):
  - Ruhr-Universitaet Bochum - St. Josef Hospital, Bochum
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitaetsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Essen Zentrum f.Kinderheilkunde Klinik f.Kinderheilkunde III, Essen
  - Universitatsklinikum Jena, Klinik fur Kinder und Jugendmedizin, Jena
  - Medizinische Klinik Innenstadt, München
  - Universitaetsklinik für Kinder- und Jugendmedizin Tuebingen, Tübingen
- Italy (11):
  - Azienda Ospedaliero Universitaria, Ospedali Riuniti, Ospedale Pediatrico G. Salesi, Ancona
  - Azienda Ospedale Policlinico di Bari, Bari
  - University of Catania, Catania
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Gastroenterologia Pediatrica E Fibrosi Cistica, Contesse -Messina
  - University Federico II of Naples, Pediatrics Department, Naples
  - Clinica di Malattie dell'Apparato Respiratorio, Orbassano (Torino)
  - Istituto Azienda Ospedaliera Universitaria, Parma
  - Universita degli Studi di Roma La Sapienza, Azienda Policlinico Umberto I, Dipartimento di Pediatria, Centro Fibrosi Cistica Regione Lazio, Roma
  - Bambino Gesu Hospital, Cystic Fibrosis Unit, Rome
  - Ospedale Infantile Regina Margherita, Turin
  - Azienda Ospedaliera Universitaria Integrata, Centro Fibrosi Cistica-Ospedale Civile Maggiore, Verona
- Poland (9):
  - Specjalistyczny Zespot Opieki Zdrowotnej nad Matka i Dzieckiem Poradnia Leczenia Mukowiscydozy, Gdansk
  - Centrum Pulmonologii i Alergologii w Karpaczu, Karpacz
  - Wojewodzki Szpital Specjalistyczny im Kopernika, Lodz
  - ALERGOTEST s.c Specjalistyczne Centrum Medyczne, Lublin
  - Szpital Kliniczny im Karola Jonschera, Poznan
  - NZOZ Sanatorium Cassia Villa Medica, Rabka-Zdrój
  - NZOZ Podkarpacki Osrodek Pulmonologii i Alergologii, Rzeszów
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - IRMED Irena Wojciechowska, Warsaw
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Sheffield Children's Hospital, The Academic Unit of Child Health, Sheffield

REFERENCES:
- [Derived] Somaraju URR, Solis-Moya A. Pancreatic enzyme replacement therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Aug 5;8(8):CD008227. doi: 10.1002/14651858.CD008227.pub4. PMID 32761612
- [Derived] Taylor CJ, Thieroff-Ekerdt R, Shiff S, Magnus L, Fleming R, Gommoll C. Comparison of two pancreatic enzyme products for exocrine insufficiency in patients with cystic fibrosis. J Cyst Fibros. 2016 Sep;15(5):675-80. doi: 10.1016/j.jcf.2016.02.010. Epub 2016 Mar 21. PMID 27013382